CLINICAL TRIAL: NCT05206994
Title: Evaluation of the Close to Home Program in California: Assessing the Impact of Community Mobilization to Prevent Sexual Violence at the Individual, Social Network, and Community Levels
Brief Title: Evaluation of the Close to Home Program in California
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California Department of Public Health (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor of Global Public Health, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201920S; U01CE003711; U01CE003201 (Other Grant/Funding Number: Centers for Disease Control and Prevention); U01CE003711 (NIH)
Record Dates: First submitted 2021-12-03; First posted 2022-01-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sexual Violence; Sexual Assault; Adolescent Behavior
Keywords: Intimate Partner Violence
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Close to Home (C2H) is a primary prevention community mobilization model that engages community members across multiple sectors and social networks to strengthen community connections and shift social norms regarding SV, but has never been rigorously evaluated. C2H moves beyond criminal justice, lobbying, or school-based curricular approaches, taking a true community-level and community-led approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Close to Home Intervention (Experimental): Sites receiving the intervention arm were determined prior to the initiation of the research. The rape crisis center in each community applied for funding from the California Department of Public Health to implement the Close to Home model in their community and they were accepted via a competitive application process. Close to Home (C2H) is a community mobilization model developed in Boston and adapted for California and is specifically designed to prevent SV by strengthening community social connections and engaging whole communities in dialogue and action to transform social norms.
  Interventions: Behavioral: Close to Home
- Control Program (No Intervention): The control program is the 4-H Youth Development Program, which is implemented across every county in California via the University of California Cooperative Extension. In 4-H programs, kids and teens complete hands-on projects in areas like health, science, agriculture and civic engagement in a positive environment where they receive guidance from adult mentors and are encouraged to take on proactive leadership roles. The model does not use community mobilization and does not address sexual violence.
  Control communities were selected based on propensity score matching using sociodemographic and community-level variables related to risk for sexual violence. The closest match was recruited first, and a next-best match was used if the first match declined participation.

INTERVENTIONS:
Behavioral: Close to Home — Close to Home (C2H), a community mobilization model developed in Boston and adapted for California, is specifically designed to prevent SV by strengthening community social connections and engaging whole communities in dialogue and action to transform social norms. The C2H model guides communities through four phases: 1) Assess, 2) Talk, 3) Build, and 4) Act. C2H mobilizes diverse groups of people residing in a shared geography and linked by social and political ties to engage in joint actions for SV prevention
  Arms: Close to Home Intervention

SUMMARY:
Investigators propose to rigorously evaluate the Close to Home (C2H) model via a cluster-matched control trial across 18 diverse communities (9 C2H, 9 control) in California via collection and analyses of social network, school-based and social media data. Close to Home is a primary prevention community mobilization model implemented in 10 communities across California that engages community members across multiple sectors and social networks to strengthen community connections and shift social norms regarding sexual violence (SV), but has never been rigorously evaluated. C2H moves beyond criminal justice, lobbying, or school-based curricular approaches, taking a true community-level and community-led approach. This is a five-year project, funded by the Centers for Disease Control and Prevention (CDC) for 3 years with competitive awards for years 4 and 5, and is conducted in partnership with the California Department of Public Health (CDPH) and ValorUs (formerly CALCASA). The University of California, San Diego (UCSD) and CDPH partnership is uniquely poised to conduct the first rigorous evaluation of C2H in California at this time.

DETAILED DESCRIPTION:
Investigators propose to rigorously evaluate the Close to Home (C2H) model via a cluster-matched control trial across 18 diverse communities (9 C2H, 9 control) in California via collection and analyses of social network, school-based and social media data. Analyses of these data will provide evidence at the individual, interpersonal and community levels of the effectiveness of this community mobilization approach to reduce sexual violence (SV) incidence. California is uniquely poised to conduct this research, given a) the multiple, diverse of communities implementing C2H; b) California Department of Public Health (CDPH)'s 10-year commitment to building capacity to support local implementation of this model, and c) CDPH's ongoing partnership on RPE evaluation with University of California San Diego's Center on Gender Equity and Health, a center with the highest levels of expertise in evaluation of SV prevention programs, and the science of social norms, social networks and social media. A Research Advisory Board will be engaged and inform and guide these efforts throughout the project period. Investigators will accomplish this highly innovative effort via the following aims:

AIM 1. Develop and implement a cluster-matched control design in partnership with the RAB, including collecting baseline social network, school-based and social media data across 14 diverse California communities.

Hypothesis 1.1: Analyses of baseline social network data will demonstrate pathways of influence regarding SV social norms and behaviors among male and female youth ages 14-24 years.

Hypothesis 1.2: Analyses of triangulated YouGov and Twitter data will yield a valid, feasible social media-based assessment of SV social norms at the community-level for evaluation of SV prevention efforts.

AIM 2: Evaluate effects of the C2H model on SV social norms and incidence, as well as patterns of diffusion of these effects, via longitudinal analyses of social network data.

Hypothesis 2.1: Social norms rejecting SV will increase, and 12-month incidence of SV will decrease at 24-month follow-up among C2H participants relative to those in control programs, and these effects will diffuse via paths of influence across social networks assessed via Aim 1.

AIM 3: Extend Aim 2 findings via analyses of multiple waves of school-based data and geocoded social media data to yield multiple tests of community-level effects of C2H on SV social norms and incidence.

Hypotheses 3.1: Analyses of data from the California Healthy Kids Survey (ages 14-19 yrs) and Twitter (>13 yrs) collected from C2H and control communities (coincident with baseline and 24-month follow-up social network data) will yield evidence of community-level effects of C2H on SV social norms and incidence consistent with individual and network-level effects observed via Aim 2 analyses.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 14-24 years old
* Must be enrolled in program with partner organization(s) or have been nominated by a peer enrolled in the partner programs
* Provide informed consent to participate

Exclusion Criteria:

* Under age 14
* Over age 24

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Virtual/Online Sexual Harassment - Digital Dating Abuse Scale | 2 years
  Two item measure sexual harassment victimization and six items measure perpetration online, over text, or through social media. Response options: yes, in the last 12 months; yes, prior to last 12 months; never. Items used are adapted from the Digital Dating Abuse Scale - Reed, L. A., Tolman, R. M., & Ward, L. M. (2017). Gender matters: Experiences and consequences of digital dating abuse victimization in adolescent dating relationships. Journal of adolescence, 59, 79-89.
In-Person Sexual Harassment & Violence - Sexual Harassment & Violence Scale | 2 years
  One item measures in-person sexual harassment victimization and three items measure perpetration. Response options: yes, in the last 12 months; yes, prior to last 12 months; never. Items were adapted from Mitchell, K. J., Ybarra, M. L., & Korchmaros, J. D. (2014). Sexual harassment among adolescents of different sexual orientations and gender identities. Child abuse & neglect, 38(2), 280-295 and Miller, E., Jones, K. A., Ripper, L., Paglisotti, T., Mulbah, P., & Abebe, K. Z. (2020). An athletic coach-delivered middle school gender violence prevention program: A cluster randomized clinical trial. JAMA pediatrics, 174(3), 241-249.
Dating Violence Victimization- Coaching Boys into Men Modified Dating Violence Victimization/Perpetration Scale | 2 years
  Two items measure dating violence victimization. Response options: yes, in the last 12 months; yes, prior to last 12 months; never. Items were adapted from Miller, E., Jones, K. A., Ripper, L., Paglisotti, T., Mulbah, P., & Abebe, K. Z. (2020). An athletic coach-delivered middle school gender violence prevention program: A cluster randomized clinical trial. JAMA pediatrics, 174(3), 241-249.
Dating Violence Perpetration- Coaching Boys into Men Modified Dating Violence Victimization/Perpetration Scale | 2 years
  Four items measure perpetration. Response options: yes, in the last 12 months; yes, prior to last 12 months; never. Items were adapted from Miller, E., Jones, K. A., Ripper, L., Paglisotti, T., Mulbah, P., & Abebe, K. Z. (2020). An athletic coach-delivered middle school gender violence prevention program: A cluster randomized clinical trial. JAMA pediatrics, 174(3), 241-249.
Sexual Violence Victimization/Perpetration - Coaching Boys into Men Modified Perpetration Scale | 2 years
  One item measures in-person sexual violence victimization and twp items measure perpetration. Response options: yes, in the last 12 months; yes, prior to last 12 months; never. Items were adapted from Miller, E., Jones, K. A., Ripper, L., Paglisotti, T., Mulbah, P., & Abebe, K. Z. (2020). An athletic coach-delivered middle school gender violence prevention program: A cluster randomized clinical trial. JAMA pediatrics, 174(3), 241-249.
LGBTQ+ and Gender Minority Violence- Victimization Scale | 2 years
  Nine items measure specific forms of sexual violence and harassment victimization experienced by sexual and gender minority youth. Response options: yes, in the last 12 months; yes, prior to last 12 months; never. Items adapted from Peitzmeier SM, Wirtz AL, Humes E. et al. The transgender-specific intimate partner violence scale for research and practice: Validation in a sample of transgender women. Social Science & Medicine. 2021. 291: 114495. https://doi.org/10.1016/j.socscimed.2021.114495 and Scheer J, Woulfe JM, Goodman LA. Psychometric validation of the identity abuse scale among LGBTQ individuals. Community Psychology. 2018.

SECONDARY OUTCOMES:
Social Norms- Sexual Violence Social Norms Scale | 2 years
  Four item scale assessing injunctive social norms related to perceived acceptability of SV among peers developed for this study; not yet validated.
Social Norms- Shared Concern about Sexual and Dating Violence Scale | 2 years
  Three item measure of social norms related to expectations of people's actions around preventing sexual and dating violence in the community (descriptive norm). Response options: 6-point Likert scale; strongly disagree to strongly agree. Adapted from Lippman 2016. Development, Validation, and Performance of a Scale to Measure Community Mobilization. Soc Sci Med. 2016 May ; 157: 127-137. doi:10.1016/j.socscimed.2016.04.002
Social Cohesion Scale | 2 years
  Two item measure of perceived social cohesion in community. Response options: 6-point Likert scale; strongly disagree to strongly agree. Items adapted from Banyard, Edwards. 2019. "What would the neighbors do?" Measuring sexual and domestic violence prevention social norms among youth and adults https://onlinelibrary.wiley.com/doi/full/10.1002/jcop.22201; Yes change: Banyard, Edwards, Rizzo 2020. Improving Social Norms and Actions to Prevent Sexual and Intimate Partner Violence: A Pilot Study of the Impact of Green Dot Community on Youth https://journals.sagepub.com/doi/full/10.1177/2632077020966571
Community Connectedness Scale | 2 years
  Four items assessing perceived connection to fellow youth in the intervention program. Response options: 6-point Likert scale; strongly disagree to strongly agree. Adapted from Lippman 2016. Development, Validation, and Performance of a Scale to Measure Community Mobilization. Soc Sci Med. 2016 May ; 157: 127-137. doi:10.1016/j.socscimed.2016.04.002
Sense of Belonging Scale | 2 years
  Two items measuring sense of belonging to the community. Response options: 6-point Likert scale; strongly disagree to strongly agree. Adapted from Fujiwara, T., & Kawachi, I. (2008). Social capital and health: a study of adult twins in the US. American journal of preventive medicine, 35(2), 139-144.
Sense of Community Scale | 2 years
  Six item scale measuring sense of community connectedness. Response options: 6-point Likert scale; strongly disagree to strongly agree. Adapted from Peterson, N.A., Speer, P.W., & Hughey, J. (2006). Measuring sense of community: A methodological interpretation of the factor structure debate. Journal of Community Psychology, 34, 453-469.

CONTACTS AND LOCATIONS:
Overall Officials: Jay G Silverman, PhD, Principal Investigator — Tulane Center on Community-Engaged GBV Research
Locations (1):
- Dr. Jay Silverman, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No